CLINICAL TRIAL: NCT01789944
Title: Peer Counseling in Family-Based Pediatric Overweight Treatment
Brief Title: Parent Partnership Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Brian Saelens, Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1R21DK095676-01 (NIH)
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Childhood Obesity
Keywords: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Provide Treatment (Experimental): Peers provide treatment to 2nd generation following receipt of the intervention.
  Interventions: Behavioral: Behavioral: Family-based behavioral intervention
- Treatment Only (Experimental): Peers receive treatment and return for a 6-month follow-up
  Interventions: Behavioral: Behavioral: Family-based behavioral intervention

INTERVENTIONS:
Behavioral: Behavioral: Family-based behavioral intervention — This behavioral treatment includes behavioral skills training and accountability, including food and activity self-monitoring, goal setting, and home environment change

SUMMARY:
To evaluate the acceptability and feasibility of peers as interventionists in delivering family-based behavioral pediatric weight control intervention.

DETAILED DESCRIPTION:
A new model of delivering family-based pediatric overweight treatment that decreases costs but sustains short- and long-term efficacy is needed. One possible opportunity for this is a peer intervention model in which families receiving professionally-led intervention then subsequently providing intervention to other families. In addition, peer interventionists' continued engagement in the behavior change process through providing intervention to others could improve their own long-term efficacy. The project begins with the standard approach of having professional interventionists provide family-based behavioral pediatric overweight treatment to overweight children and their parent (1st generation families; n=30). Subsequently, half of 1st generation families will be randomly assigned to serve as peer interventionists to other overweight parents and children (2nd generation families; n=30). The remaining 1st generation families will neither receive nor provide any additional treatment. This project aims to develop the peer intervention training and delivery and then to examine the feasibility and acceptability of the peer intervention. This project also aims to derive an estimate of the efficacy of peer intervention (receiving and providing) both at the end of receiving treatment and 6 months later, as well as the impact of providing intervention on peer interventionists' weight outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Child age: 7-11 years at time of enrollment
* Overweight child: at or above 85th percentile for age- and gender-specific BMI.
* At least one overweight parent (BMI≥ 25.0).
* Parent is willing and able to actively participate in treatment including willingness to serve as a peer interventionist following treatment.
* Must live within 50 miles of the treatment center.

Exclusion Criteria:

* Current enrollment in another weight control program for the participating child or parent.
* The participating parent is pregnant.
* Thought disorder, suicidality, or substance abuse disorder in either the participating parent or the participating child.
* Inability of the child to comprehend English at a 1st-grade level or participating parent to comprehend English at an 8th-grade level.
* Physical disability or illness in either the participating parent or the child that precludes moderate intensity physical activity.
* Medication regimen for the child that affects his or her weight.
* Conditions known to promote obesity in the participating child (e.g. Prader-Willi).
* Diagnosed eating disorder (i.e., anorexia nervosa, bulimia nervosa, binge eating disorder) in either parent (participating and nonparticipating) and/or the participating child.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Child BMI z-score | 20 Weeks

SECONDARY OUTCOMES:
Acceptability & Feasibility | 11 months
  Participant ratings based on Likert-type items regarding treatment satisfaction and helpfulness of treatment provision

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's, Seattle, Washington, United States